CLINICAL TRIAL: NCT03412643
Title: An Open-Label Phase II Trial to Evaluate the Efficacy and Safety of Neoadjuvant Doxorubicin Plus Cyclophosphamide Followed by Weekly Paclitaxel Plus Trastuzumab and Pertuzumab in Early Stage HER2-Negative Breast Cancer Patients Selected With a Test Measuring Live Cell HER2 Signaling Transduction (FACT 1)
Brief Title: Study of Neoadjuvant Chemotherapy Plus Trastuzumab and Pertuzumab in HER2-Negative Breast Cancer Patients With Abnormal HER2 Signaling
Acronym: FB-12
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Celcuity, LLC (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-12
Record Dates: First submitted 2018-01-12; First posted 2018-01-26 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: HER2-negative Breast Cancer
Keywords: NSABP; Celcuity; HER2-negative; invasive; breast cancer; Open-label; Neoadjuvant; Early stage; Doxorubicin; Cyclophosphamide; Paclitaxel; Trastuzumab; Pertuzumab; CELx HSF; HER2 Signaling Function test; anti-HER2 Antibodies
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Arm 1 (Experimental): Celcuity CELx HSF Test on tumor material obtained from research core biopsy to select patients with abnormal HER2 signaling tumors
  Doxorubicin + cyclophosphamide followed by Weekly Paclitaxel +Trastuzumab+Pertuzumab
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Weekly Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Diagnostic Test: Celcuity CELx HSF

INTERVENTIONS:
Drug: Doxorubicin — 60 mg/m2 IV Day 1 every 2 weeks or 3 weeks at investigator's discretion for a total of 4 cycles
Drug: Cyclophosphamide — 600 mg/m2 IV Day 1 every 2 weeks or 3 weeks at investigator's discretion for a total of 4 cycles
Drug: Weekly Paclitaxel — 80 mg/m2 IV weekly for 12 doses
Drug: Trastuzumab — loading dose of 8 mg/kg IV; then 6 mg/kg IV every 3 weeks for Cycles 2-4
Drug: Pertuzumab — loading dose of 840 mg IV; then 420 mg IV every 3 weeks for Cycles 2-4
Diagnostic Test: Celcuity CELx HSF — Prior to drug interventions 3, 4,and 5, the Celcuity CELx HSF diagnostic test will be conducted to assess HER2 signaling activity

SUMMARY:
This is a prospective, single arm, open label, multicenter interventional study designed to evaluate the efficacy of neoadjuvant chemotherapy with anti-HER2 antibodies in patients with HER2-negative invasive breast cancer who have abnormal HER2 signaling activity determined by the Celcuity CELx HER2 Signaling Function (HSF) testing.

DETAILED DESCRIPTION:
Patients will be required to have a prescreening research core needle biopsy to procure a fresh tumor specimen that will be sent to Celcuity for CELx HSF testing, in order to assess the status of their HER2 signaling activity (abnormally or normally active).

Patients who have abnormal HER2 signaling activity will receive weekly paclitaxel plus the anti-HER2 therapy regimen of trastuzumab and pertuzumab following completion of initial doxorubicin/cyclophosphamide.The primary endpoint of the study is to evaluate whether patients with HER2-negative breast cancers based on standard American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) testing criteria, but with abnormal HER2-driven signaling pathways determined by the Celcuity HSF assay and receive HER2-targeted therapy with neoadjuvant chemotherapy, will have a higher rate of pathological complete response in the breast and lymph nodes (pCR breast and lymph nodes) than has been found historically in patients with HER2-negative breast cancer who have received neoadjuvant chemotherapy alone. Secondary endpoints include pathologic complete response (breast), clinical complete response (cCR), residual cancer burden (RCB) 0-1 index, and relationship between quantitative CELx score and pCR rate.

It is expected that approximately 270 patients will need to be prescreened in order to enroll 54 patients (26 ER-positive/HER2-negative and 28 ER-negative/HER2-negative) who have abnormal HER2 signaling activity.

ELIGIBILITY:
Inclusion Criteria:

SCREENING PRIOR TO INITIATING CHEMOTHERAPY

Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy.

The primary breast tumor must be palpable and measure greater than or equal 2.0 cm on physical exam.

The regional lymph nodes can be cN0, cN1, or cN2a.

Histological grade II or III tumor.

Ipsilateral axillary lymph nodes must be evaluated by imaging (mammogram, ultrasound, and/or MRI) within 6 weeks prior to initiating chemotherapy. If suspicious or abnormal, FNA or core biopsy is recommended, also within 6 weeks prior to initiating chemotherapy. Findings of these evaluations will be used to determine the nodal status prior to initiating chemotherapy.

* Nodal status - negative: Imaging of the axilla is negative; Imaging is suspicious or abnormal but the FNA or core biopsy of the questionable node(s) on imaging is negative;
* Nodal status - positive: FNA or core biopsy of the node(s) is cytologically or histologically suspicious or positive. Imaging is suspicious or abnormal but FNA or core biopsy was not performed.

Tumor specimen obtained at the time of diagnosis must have ER and progesterone receptor (PgR) analysis assessed by current ASCO/CAP Guidelines. Patients are eligible with either hormone receptor-positive or hormone receptor-negative tumors.

Tumor specimen obtained at the time of diagnosis must have been determined to be HER2-negative as follows:

* Immunohistochemistry (IHC) 0-1+; or
* IHC 2+ and in situ hybridization (ISH) non-amplified with a ratio of HER2 to chromosome enumeration probe 17 (CEP17) less than 2.0, and if reported, average HER2 gene copy number less than 4 signals/cells; or
* ISH non-amplified with a ratio of HER2 to CEP17 less than 2.0, and if reported, average HER2 gene copy number less than 4 signals/cells.

Blood counts performed within 6 weeks prior to initiating chemotherapy must meet the following criteria:

* absolute neutrophil count (ANC) must be greater than or equal 1200/mm3;
* platelet count must be greater than or equal 100,000/mm3; and
* hemoglobin must be greater than or equal 10 g/dL.

The following criteria for evidence of adequate hepatic function performed within 6 weeks prior to initiating chemotherapy must be met:

* total bilirubin must be less than or equal to upper limit of normal (ULN) for the lab unless the patient has a bilirubin elevation greater than ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
* alkaline phosphatase must be less than or equal to 2.5 x ULN for the lab; and
* aspartate aminotransferase (AST) must be less than or equal to 1.5 x ULN for the lab.
* Alkaline phosphatase and AST may not both be greater than the ULN. For example, if the alkaline phosphatase is greater than the ULN but less than or equal to 2.5 x ULN, the AST must be less than or equal to the ULN. If the AST is greater than the ULN but less than or equal to 1.5 x ULN, the alkaline phosphatase must be less than or equal to ULN. Note: If alanine aminotransferase (ALT) is performed instead of AST (per institution's standard practice), the ALT value must be less than or equal to 1.5 x ULN; if both were performed, the AST must be less than or equal to 1.5 x ULN.

Patients with AST or alkaline phosphatase greater than ULN are eligible for inclusion in the study if liver imaging (CT, MRI, PET-CT, or PET scan) performed within 6 weeks prior to initiating chemotherapy does not demonstrate metastatic disease and the requirements in next criteria are met.

Patients with alkaline phosphatase that is greater than ULN but less than or equal to 2.5 x ULN or unexplained bone pain are eligible for inclusion in the study if a bone scan, PET-CT scan, or positron emission tomography (PET) scan performed within 6 weeks prior to initiating chemotherapy does not demonstrate metastatic disease.

Serum creatinine performed within 6 weeks prior to initiating chemotherapy must be less than or equal to 1.5 x ULN for the lab.

The left ventricular ejection fraction (LVEF) assessment by echocardiogram or multi-gated acquisition (MUGA) scan performed within 90 days prior to initiating chemotherapy must be greater than or equal 55 percent regardless of the facility's lower limit of normal (LLN).

Patients with reproductive potential must agree to use an effective non-hormonal method of contraception during therapy and for at least 7 months after the last dose of study

MAIN STUDY ENROLLMENT

Tumor determined to have abnormal HER2-driven signaling activity based on the CELx HSF test.

______________

Exclusion Criteria:

T4 tumors including inflammatory breast cancer.

FNA alone to diagnose the breast cancer.

Excisional biopsy or lumpectomy performed prior to initiating chemotherapy.

Surgical axillary staging procedure prior to initiating chemotherapy. Pre-neoadjuvant therapy sentinel node biopsy is not permitted. (FNA or core biopsy is acceptable.)

Definitive clinical or radiologic evidence of metastatic disease. Required imaging studies must have been performed within 6 weeks prior to initiating chemotherapy.

Synchronous bilateral invasive breast cancer. (Patients with synchronous and/or previous contralateral ductal carcinoma in situ [DCIS] or lobular carcinoma in situ [LCIS] are eligible.)

Any previous history of ipsilateral invasive breast cancer or ipsilateral DCIS. (Patients with synchronous or previous ipsilateral LCIS are eligible.)

Previous therapy with anthracycline, taxanes, trastuzumab, or other HER2 targeted therapies for any malignancy.

Any sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy, etc. (These patients are eligible if this therapy is discontinued prior to initiating chemotherapy.)

History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 2 years prior to initiating chemotherapy.

Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimens. This includes but is not confined to:

* Active cardiac disease: angina pectoris that requires the use of anti-anginal medication; ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; valvular disease with documented compromise in cardiac function; and symptomatic pericarditis.
* History of cardiac disease: myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular (LV) function; history of documented congestive heart failure (CHF); and documented cardiomyopathy.

Uncontrolled hypertension defined as sustained systolic BP greater than 150 mmHg or diastolic BP greater than 90 mmHg. (Patients with initial BP elevations are eligible prior to initiating chemotherapy if initiation or adjustment of BP medication lowers pressure.)

Active hepatitis B or hepatitis C with abnormal liver function tests. Intrinsic lung disease resulting in dyspnea.

Poorly controlled diabetes mellitus.

Active infection or chronic infection requiring chronic suppressive antibiotics.

Patients known to be HIV positive.

Nervous system disorder (paresthesia, peripheral motor neuropathy, or peripheral sensory neuropathy) greater than or equal to grade 2, per the CTCAE v4.0.

Malabsorption syndrome, ulcerative colitis, resection of the stomach or small bowel, or other disease significantly affecting gastrointestinal function.

Other non-malignant systemic disease that would preclude treatment with any of the treatment regimens or would prevent required follow-up.

Conditions that would prohibit administration of corticosteroids.

Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids).

Known hypersensitivity to any of the study drugs or any of the ingredients or excipients of these drugs (e.g., Cremophor EL), including sensitivity to benzyl alcohol.

Pregnancy or lactation at the initiation of chemotherapy. (Note: Pregnancy testing must be performed within 2 weeks prior to initiating chemotherapy according to institutional standards for women of childbearing potential.)

Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (PCR) to study therapy (both breast and lymph node-combined; ypT0/Tis ypN0) | From initiation of study therapy to time of surgery, which is usually performed 3 to 4 weeks after completion of study therapy
  Percentage of patients with absence of residual invasive cancer in H&E slides of resected breast specimens and all sampled regional lymph nodes following the completion of neoadjuvant systemic therapy

SECONDARY OUTCOMES:
Pathologic complete response to study therapy (breast) | From initiation of study therapy to time of surgery, which is usually performed 3 to 4 weeks after completion of study therapy
  Percentage of patients with absence of residual invasive cancer in H&E slides of resected breast specimens following the completion of neoadjuvant systemic therapy
Clinical complete response (both breast and axilla) | From initiation of study therapy to 2-4 weeks after completion of study therapy
  Percentage of patients with clinical complete response (cCR) measured by physical examination of the breast and axilla
Residual cancer burden (RCB) | From initiation of study therapy to time of surgery, which is usually performed 3 to 4 weeks after completion of study therapy
  Combined index of pathologic measurements of residual tumor size and cellularity and number and size of regional lymph nodes
Logistic regression | From prior to study entry (time of CELx score assay) to 4-6 weeks after surgery (pCR outcome determination)
  Regression of quantitative CELx scores by pCR outcome
Frequency of adverse events assessed by CTCAE 4.0 | From beginning of study therapy to 4-6 weeks after surgery
  Frequency of adverse events categorized using the NCI Common Terminology Criteria for Adverse Events version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (43):
- United States (43):
  - Arrowhead Regional Medical Center, Colton, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University of Florida Cancer Center at Orlando Health, Orlando, Florida
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Louisville JG Brown Cancer Center, Louisville, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Herbert Herman Cancer Center, Sparrow Hospital, Lansing, Michigan
  - Ascension St. Mary's, Saginaw, Michigan
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of Rochester - Wilmot Cancer Institute, Rochester, New York
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Hospital, Canton, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital & Richard Solove Research Institute, Columbus, Ohio
  - Columbus Oncology & Hematology Associates Inc, Columbus, Ohio
  - The Mark H. Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Adena Regional Medical Center, Columbus, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Dayton Physicians LLC, Dayton, Ohio
  - Delaware Health Center, Delaware, Ohio
  - Marietta Memorial Hospital Cancer Center, Marietta, Ohio
  - Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Genesis Health Care, Zanesville, Ohio
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - Harris Health Systems-Smith Clinic, Houston, Texas
  - Lester and Sue Smith Breast Center, Houston, Texas
  - Centra Lynchburg Hematology Oncology, Lynchburg, Virginia
  - Bon Secours Richmond Community Hospital Medical Oncology Assoc., Mechanicsville, Virginia
  - Bon Secours St. Francis Medical Center, Midlothian, Virginia
  - Bon Secours Richmond Community Hospital at St. Mary's, Richmond, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Ascension St. Elizabeth Hospital, Appleton, Wisconsin